CLINICAL TRIAL: NCT03272828
Title: A Prospective Randomized Study on the Immediate Loading of Mandibular Overdentures Supported by Parallel Sided or Tapered Dental Titanium Implants
Brief Title: Mandibular Overdenture Clinical Trial Comparing Parallel Sided and Tapered Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Mats Kronstrom, Professor, Department of Restorative Dentistry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003063
Record Dates: First submitted 2017-09-02; First posted 2017-09-06 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Parallel sided implant Group (Active Comparator): A Parallel sided titanium dental implant will be placed in the edentulous mandible.
  Interventions: Device: Nobel Biocare titanium dental implants
- Tapered shaped implant Group (Active Comparator): A tapered shaped titanium dental implant will be placed in the edentulous mandible.
  Interventions: Device: Nobel Biocare titanium dental implants

INTERVENTIONS:
Device: Nobel Biocare titanium dental implants

SUMMARY:
The purpose of the study is to compare two different types of dental implants which will be used to support/retain a removable denture in the edentulous mandible. Subjects will have one implant placed in the midline of the mandible after which the patient's existing denture will be modified to fit the implant. The population of this study consists of healthy edentulous individuals 20-75 years of age who have complete dentures in the upper and lower arch.

DETAILED DESCRIPTION:
Titanium dental implants have been frequently used in the rehabilitation of edentulous patients. Implants may provide adequate denture stability, improve oral function and oral health related quality of life. There is evidence that implants supporting fixed and removable prostheses have excellent long term success rates. Factors such as implant surface characteristics, length, diameter and shape (parallel sided or tapered) may play and important role for the outcome of the treatment especially when the immediate loading protocol (loading of the implant the same day it is surgically placed) is utilized. There are reports indicating that dental implants placed according to the immediate loading protocol can be used to support removable prostheses in the mandible. Such protocol would minimize the number of surgical procedures and significantly shorten the overall treatment time. Further, increased oral health related quality of life has been reported from studies on mandibular implant overdentures. Traditionally two implants have been suggested for the support of a mandibular overdenture. However, high patient satisfaction rates and appropriate denture retention have been reported among patients with a single implant placed in the mid-line. It is also important to further evaluate and compare various implant designs to determine clinical outcomes. The two dominating types of implant body design on the market are the parallel-sided (straight) and the tapered (conical) shaped. Both implants have similar threads, and the surgical procedure for placing the implants in the bone tissue is similar, but the drills used have a slightly different design and shape. There are today no randomized controlled studies evaluating differences in outcomes with respect to the external implant design i.e. parallel sided or tapered.

ELIGIBILITY:
Inclusion Criteria:

* Be between 20 and 75 years of age
* Be edentulous and have both upper and lower complete dentures
* Present with American Society of Anesthesiologists (ASA) I or ASA II and no medical contraindications to implant treatment
* Have adequate bone volume for placement of one (1) 4.0 mm diameter titanium dental implant with a minimum length of 10 mm in the symphyseal area (=midline) of the anterior mandible
* Show absence of pathology such as cysts, infections in the gum tissue or bone and remaining roots.
* Be able to understand the procedures and have a jaw opening range of 30 mm or more

Exclusion Criteria:

* Ongoing chemotherapy
* Previous radiation to head/neck
* Ongoing corticosteroid medication
* Ongoing blood thinner medication
* Ongoing medication with psychopharmacological drugs
* History of alcohol/drug abuse
* Remaining teeth/root tips
* Poor quality /fractured/severely worn dentures that cannot be modified to fit the implant
* Jaw opening range less than 30 mm

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mats Kronstrom, DDS, PhD, Principal Investigator — University of Washington
Locations (1):
- the Regional Research Clinic, School of Dentistry at the University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with other researchers

REFERENCES:
- [Background] Kronstrom M, Davis B, Loney R, Gerrow J, Hollender L. Satisfaction and Clinical Outcomes Among Patients with Immediately Loaded Mandibular Overdentures Supported by One or Two Dental Implants: Results of a 5-Year Prospective Randomized Clinical Trial. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):128-136. doi: 10.11607/jomi.4824. PMID 28095527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via flyers posted in the School of Dentistry. A total of 63 people were screened for eligibility and 48 met the inclusion criteria.
Pre-assignment Details: Of 48 eligible participants who signed the consent form and were enrolled in the study, one declined study participation due to lack of willingness to pay for the required cone beam computed tomography (CBCT) pre-surgical procedure. Participants were randomized to implant group the day of surgery.
Groups:
- Parallel Sided Implant Group: A Parallel sided titanium dental implant will be placed in the edentulous mandible.
  Nobel Biocare titanium dental implants
- Tapered Shaped Implant Group: A tapered shaped titanium dental implant will be placed in the edentulous mandible.
  Nobel Biocare titanium dental implants
Period: Overall Study
Arm/Group | Parallel Sided Implant Group | Tapered Shaped Implant Group
Started | 24 | 23
Completed | 13 | 13
Not Completed | 11 | 10
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Deceased | 1 | 1
Not completed — Failed implant | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parallel Sided Implant Group | Tapered Shaped Implant Group | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Full Range); unit: years] | 61.17 [43 to 74] | 61.74 [43 to 75] | 61.45 [43 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 9 | 12 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 23 | 47
Implant stability quotient (ISQ) [Mean (Standard Deviation); unit: units on a scale] — The ISQ is obtained by resonance frequency measurement after an implant is placed. The value of the measurement ranges from 1 to 100 with higher values indicating greater stability.
  units on a scale | 82.75 (2.75) | 81.30 (3.65) | 82.04 (3.27)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Implant Failure Rate Between Parallel Sided and Tapered Dental Implants at 5 Years
Description: Implant failure defined as an implant that has lost osseointegration and no longer is stable and supported by the surrounding bone (no bone to implant contact).
Time Frame: From implant placement (baseline) to 5 years
Population: All participants who had an implant placed at the midline of the mandibular arch and their mandibular denture fitted for immediate wearing.
Measure: Count of Participants; unit: Participants
Arm/Group | Parallel Sided Implant Group | Tapered Shaped Implant Group
Number analyzed (Participants) | 24 | 23
Participants | 1 | 2
Statistical Analysis 1: Comparison: Parallel Sided Implant Group vs Tapered Shaped Implant Group; Test type: Superiority; p = 0.63, Fisher Exact

2. Secondary Outcome: Implant Stability Quotient (ISQ) Measured at 5 Years
Description: The implant stability quotient (ISQ) value is a measurement of the mechanical implant stability in the bone and is measured directly after surgical implant placement and then at follow-ups. It is obtained by resonance frequency with a device that sends out a signal to a metal rod placed in the implant and then reads the value of the signal when it bounces back. The value ranges from 0 to 100 with higher values indicating better bone-to-implant contact and greater stability.
Time Frame: 5 years
Population: Participants continuing in the study at 5 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parallel Sided Implant Group | Tapered Shaped Implant Group
Number analyzed (Participants) | 13 | 13
units on a scale | 80.77 (5.82) | 85.54 (6.50)
Statistical Analysis 1: Comparison: Parallel Sided Implant Group vs Tapered Shaped Implant Group; Test type: Superiority; p = 0.06, Unequal-variance 2-sample t-test

3. Secondary Outcome: Bone Loss Measurement at 5 Years
Description: The measure of bone loss in millimeters (mm) around the implant at 5 years compared to bone height at baseline. Changes in bone level are measured on intraoral radiographs and compared with the bone level measure immediately after surgical implant placement (baseline). The implant platform was used as the reference point and measurements of the bone were made to the nearest thread. The bone level is measured on both sides (mesial & distal) of the implant using the thread on the implant as reference. The distance between the threads is 0.6 mm.
Time Frame: From implant placement (baseline) to 5 years
Population: Participants continuing in the study at 5 years
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Parallel Sided Implant Group | Tapered Shaped Implant Group
Number analyzed (Participants) | 13 | 13
millimeters | 1.02 (1.37) | 0.65 (1.08)
Statistical Analysis 1: Comparison: Parallel Sided Implant Group vs Tapered Shaped Implant Group; Test type: Superiority; p = 0.45, Unequal-variance 2-sample t-test

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Parallel Sided Implant Group | Tapered Shaped Implant Group
All-Cause Mortality (participants affected / at risk) | 1/24 | 1/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 2/24 | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Parallel Sided Implant Group (N=24) | Tapered Shaped Implant Group (N=23)
Implant failure (Gastrointestinal disorders) | 1 | 2
Participant wanted implant removed (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-05-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT03272828/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT03272828/SAP_001.pdf